CLINICAL TRIAL: NCT05337371
Title: Incidence of Early Cardiac Arrythmias Following Hospital Discharge After Cardiac Arrest Monitored With Philips ePatch® 2.0
Brief Title: Cardiac Arrest Post-Discharge ECG Monitoring
Acronym: CArPEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Tharusan Thevathasan, Dr., Charite University, Berlin, Germany
Other Study IDs: Cardiac Arrest ECG
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Heart Arrest; Arrhythmias, Cardiac; Electrocardiography
MeSH Terms: conditions — Heart Arrest; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Philips ePatch® 2.0: Patients who are discharged from the hospital with ECG patch (Philips ePatch® 2.0).
  Interventions: Device: ECG patch (Philips ePatch® 2.0)

INTERVENTIONS:
Device: ECG patch (Philips ePatch® 2.0) — The ECG patch will be put on the patients chest to monitor cardiac activity for a total time period of 14 days after cardiac arrest.

SUMMARY:
The primary aim is to conduct a prospective observational cohort study to analyze the incidence of serious arrhythmic events that occur within 14 days after hospital discharge in patients who had been hospitalized for cardiac arrest caused by acute myocardial infarction. Cardiac arrythmias following hospital dischagre will be detected with Philips ePatch® 2.0 for 14 days.

DETAILED DESCRIPTION:
Approximately 60,000 patients suffer from out-of-hospital cardiac arrest in Germany every year. Areas of myocardial ischemia may induce cardiac arrythmias, such as atrial fibrillation, ventricular tachycardia or ventricular fibrillation, which are known arrhythmic complications following cardiac arrest. Additionally, an imbalance in electrolytes as well as an increased use of inotropic or vasoactive medication as part of post-resuscitation care in the intensive care unit (ICU) may further increase the risk of cardiac arrythmias. 80% of cardiac arrythmias occur within 24 hours after cardiac arrest in the ICU. Patients with cardiac arrythmias following cardiac arrest have an increased mortality risk. Therefore, patients with cardiac arrest are monitored closely with telemetric monitors in the hospital, revascularized early and treated with beta-blockers, statins and renin-angiotensin-aldosterone antagonists to enhance myocardial remodeling and to decrease the rate of cardiac arrythmias. As soon as the patients are discharged from the hospital, no telemetric ECG monitoring can be provided. Therefore, the incidence of early cardiac arrythmias, which occur within 14 days after hospital discharge after treatment for cardiac arrest, remains unclear.

We plan to include 100 adult patients (≥18 years and ≤80 years) who survived cardiac arrest caused by acute myocardial infarction within the past 10 days. Patients with a left-ventricular ejection fraction between 36 to 50% and with sinus rhythm at the time of hospital discharge will be enrolled in this study. Patients who are suitable for implantable cardioverter-defibrillators (ICD) or pacemakers, with known paroxysmal or persistent atrial fibrillation, known inability to comply with follow-up or known pregnancy will not be enrolled.

Primary aim: The primary aim is to conduct a prospective observational cohort study to analyze the incidence of serious arrhythmic events that occur within 14 days after hospital discharge in patients who had been hospitalized for cardiac arrest caused by acute myocardial infarction. Cardiac arrythmias following hospital dischagre will be detected with Philips ePatch® 2.0 for 14 days.

Secondary aims: The secondary aim is to analzye the incidence of sinus arrest, atrial fibrillation, higher degree AV-block, ventricular tachycardia or fibrillation, all-cause mortality, cardiovascular mortality, stroke, systemic arterial thromboembolism and unplanned hospitalizations for decompensated heart failure within 14 days after discharge from the index hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years
* Cardiac arrest due to acute myocardial infarction
* Cardiac arrest ≤10 days ago
* Left-ventricular ejecion fraction at hospital discharge: 36-50%
* Sinus rhythm at hospital discharge
* Optimal medical therapy

Exclusion Criteria:

* Non-adult patients
* Cardiac arrest due to another cause other than acute myocardial infarction
* Philips ePatch® 2.0 not applicable
* ICD or pacemaker indication
* Known paroxysmal or persistent atrial fibrillation
* Inability to comply with follow-up- Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to include adult patients who survived cardiac arrest caused by acute myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious cardiac arrythmias | Cardiac arrythmias within 14 days after hospital discharge from index hospital stay following cardiac arrest event.
  Cardiac arrythmias monitored with Philips ePatch 2.0

SECONDARY OUTCOMES:
Incidence of sinus arrest, atrial fibrillation, higher degree AV-block, ventricular tachycardia or fibrillation | Cardiac arrythmias within 14 days after hospital discharge from index hospital stay following cardiac arrest event.
  Cardiac arrythmias monitored with Philips ePatch 2.0
All-cause mortality | Mortality due to any cause within 14 days after hospital discharge from index hospital stay following cardiac arrest event.
  Mortality due to any cause
Cardiovascular mortality | Mortality due to a cardiavascular cause within 14 days after hospital discharge from index hospital stay following cardiac arrest event.
  Mortality due to a cardiavascular cause
Stroke | Stroke within 14 days after hospital discharge from index hospital stay following cardiac arrest event.
  Incidence of stroke
Systemic arterial thromboembolism | Systemic arterial thromboembolism within 14 days after hospital discharge from index hospital stay following cardiac arrest event.
  Incidence of systemic arterial thromboembolism
Unplanned hospitalizations for decompensated heart failure | Unplanned hospitalizations for decompensated heart failure within 14 days after hospital discharge from index hospital stay following cardiac arrest event.
  Unplanned hospitalizations for decompensated heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skurk, MD, Study Director — Charité - University Hospital Berlin; Tharusan Thevathasan, MD, Principal Investigator — Charité - University Hospital Berlin

IPD SHARING:
Plan to Share IPD: No